CLINICAL TRIAL: NCT04721236
Title: COVID-19 Wave II Study for Assessing the Early Use of Hyperimmune Plasma for the Treatment of COVID-19 Patients Needing Non-invasive or Invasive Mechanical Ventilation
Brief Title: Early Use of Hyperimmune Plasma in COVID-19
Acronym: COV-II-PLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catherine Klersy (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor-Investigator, Catherine Klersy, Study Statistician, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100490/2020
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: hyperimmune plasma; positive pressure respiratory support
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: a multiple center, one arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): hyperimmune plasma with titre 1:80 or more
  Interventions: Other: hyperimmune plasma

INTERVENTIONS:
Other: hyperimmune plasma — plasma collected from convalescent Covid-19 donors with titre 1:80 or more

SUMMARY:
The study assesses the efficacy of early administration of hyperimmune plasma in covid-19 patients who are on CPAP or intubated. Efficacy is measured as a 2 point decrease in the WHO scale

DETAILED DESCRIPTION:
Patients who satisfy eligibility criteria and in particular have started positive pressure respiratory support not more than no more than 48 hours are administered 200 to 300 ml in 2 or 3 times administered over a time window of 5 days. . Plasma titration will depend on the availability in the local Plasma Bank; any titre ≥ 1:80 will be acceptable. primary endpoint will be assessed at 28 days; vital status will be further investigated at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performing study procedures. Witnessed oral consent will be accepted in order to avoid paper handling. Written consent by patient or representatives will be obtained as soon as possible.
2. Male or female adult patient ≥18 years of age at time of enrolment.
3. Laboratory-confirmed SARS-CoV-2 infection as determined by real-time RT-PCR in naso/oropharyngeal swabs or any other relevant specimen..
4. Patient is hospitalized for COVID-19, is severely hypoxic with a P/F ≤ 200 while breathing room air or supplemental oxygen and requires positive pressure respiratory support, either non-invasive (helmet/mask CPAP or NIV) or invasive (endotracheal intubation and mechanical ventilation)
5. No more than 48 hours between the onset of positive pressure respiratory support and treatment administration day
6. Evidence of pulmonary infiltrates at chest imaging (chest x-ray, CT scan or LUS)
7. The patient is not eligible in the Tsunami trial.

Exclusion Criteria:

1. Participation in any other clinical trial of an experimental treatment for COVID-19.
2. In the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
3. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR <30).
4. Pregnancy
5. Current documented and uncontrolled bacterial infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2022-05-19 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement (efficacy) | 28 days
  Clinical improvement is obtained when a patient decreases his/her score by 2 points on the ten-category ordinal WHO scale or is discharged alive from the hospital, whichever comes first. The WHO scale is chosen in accordance with the "Clinical Characterisation and Management Working Group of the WHO Research and Development Blueprint programme" recently published in Lancet Infectious Diseases (WHO, 2020).

SECONDARY OUTCOMES:
ventilation | Days: from 0 to 7, 14 and 28
  Ventilator-free days
WHO (World Health Organization) scale | From day 0 to 28 days
  WHO scale score reached. Minimum score is 0: unifected (no viral RNA detected); maximum score 10 (dead)
SOFA (Sequential Organ Failure Assessment) score | Days: from 0 to 7, 14 and 28
  Sequential Organ Failure Assessment Score (SOFA score). This score is used to determine the extent of a person's organ function or rate of failure, from 0 to 24, with severity increasing with higher the scores
naso-pharyngeal swab | Days: from 0 to 7, 14 and 28
  Time to a negative SARS-COV2 naso-pharyngeal swab for upper respiratory tract or BAL/BRASP for lower respiratory
SARS-CoV2 | 28 days
  Log10 change in SARS-CoV2
P/F | Days: from 0 to 7, 14 and 28
  P/F ratio. P/F is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage)
thrombosis | Days: from 0 to 7, 14 and 28
  Occurrence of deep vein thrombosis or pulmonary embolism assessed using the most appropriate imaging approach
curarization | Days: from 0 to 7, 14 and 28
  Total duration of mechanical ventilation, ventilatory weaning and curarisation in days
complication kidney | Days: from 0 to 7, 14 and 28
  KDIGO score Kidney Disease: Improving Global Outcomes (KDIGO)
complication lung | Days: from 0 to 7, 14 and 28
  Occurrence of ventilator-acquired pneumonia - Radiological and clinical context associated with a bacteriological sampling in culture of tracheal secretions, bronchiolar-alveolar lavage or a protected distal sampling
Leucocytes | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: Leucocytes (x10^3/ul)
Lymphocytes | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: Lymphocytes (x10^3/ul)
C-reactive protein | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: C-reactive protein (mg/dL)
D-dimer | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: D-dimer (ug/L)
Troponin I (TnI) | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: TNI (ng/L)
PCTI (Procalcitonin) (ng/mL) | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: PCTI (Procalcitonin) (ng/mL)
Ferritin | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: Ferritin (ng/ml)
Albumin | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: Albumin (mg/dL)
LDH | Days: from 0 to 7, 14 and 28
  Biological efficacy endpoints: LDH (mU/mL)
Lung Ultrasound Score (LUS) | Days: from 0 to 7, 14 , 28 and 6 months
  Total Lung Ultrasound Score S score
ecmo | 28 days
  Occurrence of ECMO implant
death | 28 days, 3 and 6 months
  All cause mortality
hospitalization | 28 days
  days total hospitalization and of ICU hospitalization
Lung Function tests | 6 months
  Lung Function tests
High resolution computed tomography (HRCT) | 6 months
  HRCT findings of the thorax
Improvement mortality | 28 days
  rate of clinical improvement and mortality between the patients in the study and the cohort enrolled in the local SMACORE registry

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mojoli, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Catherine Klersy, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
may be available upon motivated requesto to PI